CLINICAL TRIAL: NCT01912794
Title: Postural Responses to External Perturbation in Post-Stroke: Sensorimotor Integration and Rehabilitation
Brief Title: Postural Responses to External Perturbation in Post-Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Alessandra Rezende Martinelli, PhD student, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMH-2011/18173-3
Record Dates: First submitted 2013-07-26; First posted 2013-07-31 (Estimated); Last update posted 2013-08-01 (Estimated); Status verified 2013-07

CONDITIONS: Stroke
Keywords: Cerebrovascular Accident; Rehabilitation; Sensory System
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sensory Conditions (Experimental)
  Interventions: Other: Sensory Intervention

INTERVENTIONS:
Other: Sensory Intervention — 1. full sensory information, whose participants will practice balancing tasks without constraint sensory body;
  2. sensory constraint, whose participants will practice the same balance tasks with constraint body of visual and tactile information from the soles of the feet;
  3. control, whose participants will exercise activities involving cognitive and upper limbs.

SUMMARY:
To maintain stable body balance in daily activities, the ability to respond to external perturbations is an essential factor. Such capacity is limited in pathological conditions, such as in stroke, in which postural control is impaired due to lesions to the central nervous system. Impairment to postural control increases body sway during upright posture and leads to augmented frequency of falls. In this sense, the identification of mechanisms involved in body balance disorders after stroke is particularly important in situations of postural perturbation. The purpose of this project is to evaluate reactive postural responses to unpredictable external perturbations, analyzing postural dysfunctions caused by lesion to different brain areas as a result of stroke, and test principles of dynamic body balance rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria are as follows. Healthy participants: absence of detectable neurological or physical malfunction which might affect postural control, no use of drugs affecting body balance and preserved mental capacity. Stroke patients: capacity to sustain independently orthostatic posture for at least 5 min. and preserved mental capacity.

Exclusion Criteria:

* Exclusion Criteria are: no orthopedic malfunction, no clinical instability associated with systemic disease, no use of drugs affecting body balance and presence of "pusher syndrome".

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-02 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Displacement amplitude of the CP to the anterior-posterior and medial-lateral | 2 months
  This outcome measure quantified by the difference between the maximum values of the anterior-posterior and medial-lateral after the start of trial and average position in the axis anteroposterior and mediolateral, respectively, in the 200 ms prior to the onset of the trial.

SECONDARY OUTCOMES:
Coordination between the hip and ankle joint | 2 months
  Coordination between the hip and ankle joints, which is evaluated by adjusting the angle displacement data, hip and ankle angle within 95% of an ellipse surrounding the values of the disturbance moment until the end of the trial. Will be carried out a regression analysis to identify the slope of the fitted ellipse. Slopes greater indicate a greater share of the ankle in relation to the hip

OTHER OUTCOMES:
Muscle activation latency | 2 months
  This outcome measure is time between the time of release and the first load value 3 standard deviations above the mean magnitude in the 200 ms prior to postural disturbance, with subsequent values increasing.

CONTACTS AND LOCATIONS:
Overall Officials: Luis A Teixeira, PhD, Study Director
Locations (1):
- Escola de Educação física e Esporte, Universidade de São Paulo, São Paulo, São Paulo, Brazil